CLINICAL TRIAL: NCT04904445
Title: COVID-19 Antibody Responses In Cystic Fibrosis
Acronym: CAR-CF
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Queen's University, Belfast (Other); Cystic Fibrosis Foundation (Other); European Cystic Fibrosis Society - Clinical Trials Network (Other)
Responsible Party: Principal Investigator, Hettie M Janssens, MD PhD, Pediatric Pulmonologist, Erasmus Medical Center
Other Study IDs: NL
Record Dates: First submitted 2021-05-17; First posted 2021-05-27 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; COVID-19; SARS-CoV-2; Seroprevalence
MeSH Terms: conditions — Cystic Fibrosis; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A 6-monthly blood sample will be collected when the participants attend clinic or hospital.
  For participants who consent to the optional study, a second blood sample will also be drawn.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Coronavirus disease 2019 (COVID-19) which is caused by the virus SARS-CoV-2 has resulted in an ongoing global pandemic. It is unclear whether the relatively low number of reported cases of COVID-19 in people with CF (pwCF) is due to enhanced infection prevention practices or whether pwCF have protective genetic/immune factors. This study aims to prospectively assess the proportion of pwCF, including both adults and children with CF who have evidence of SARS-CoV-2 antibodies over a two-year period. This study will also examine whether pwCF who have antibodies for SARS-CoV-2 have a different clinical presentation and what impact this has on their CF disease. The proposed study will recruit pwCF from paediatric and adult CF centres throughout the United Kingdom. Serological testing to detect antibodies will be performed on blood samples taken at month 0, 6, 12, 18 and 24 with additional time-points if bloodwork is available via normal clinical care. Clinical data on, lung function, CF-related medical history, pulmonary exacerbations, antibiotic use, and microbiology and vaccination receipt, will be collected during routine clinical assessments.

Associations will be examined between socio-demographic and clinical variables and serologic testing. The effects of SARS-CoV-2 infection on clinical outcomes and analyse end-points will be examined to explore any age-related or gender-based differences, as well as subgroup analysis of outcomes in lung-transplant recipients and pwCF receiving CFTR modulator therapies. As pwCF receive COVID-19 vaccination a comparison of the development and progression of anti-SARS-CoV-2 antibodies in pwCF following natural infection and vaccination SARS-CoV-2 over time will be performed.

DETAILED DESCRIPTION:
This is a prospective, longitudinal cohort study in people with Cystic Fibrosis (pwCF) that involves repeated serial sampling of participants. This study design was chosen to provide comprehensive information on SARS-CoV-2 seroprevalence changes over time and the subsequent clinical impact on pwCF. The study will be conducted at participating CF centres over a 3-year period. Study participants will include paediatric and adult pwCF. Participating investigators can enrol all eligible pwCF over a 12-month period. Participants are then followed up for 24 months. Participants will donate blood samples at their routine clinic visits. Blood samples will be collected at Day 0 (baseline), at Months 6, 12, 18 and 24 (to coincide with routine clinical reviews). Additional blood samples will be taken opportunistically every time the participant visits the clinic for blood draws. These blood samples could be related to, routine care, annual review visits, pulmonary exacerbations (PEx), CF complications or when initiating new treatments (e.g. CFTR modulators).

Serum from blood samples will be shipped to a central laboratory (Queen's University Belfast) for standardized measurement of SARS-CoV-2 antibodies.

Alongside the blood samples the investigator will also collect clinical data from the patient's health records and will input this data into the case report form (CRF). Clinical data will be collected in conjunction with routine care visits, according to local clinical practice. Investigators will collect data elements from information routinely recorded in the patients' medical records. Data will be collected at baseline, month 6, 12, 18 and 24 as per the study schedule, and at additional blood sampling timepoints as previously explained above. Data collection will include routine data available from CF clinic follow-ups including background demographic information, CF medical history, medications, exacerbation information, sputum microbiology and clinical and lung function parameters. Information on SARS-CoV-2 infection history and vaccine receipt will also be collected.

The maximum follow-up duration of participation in the study for each patient will be 24 months. This study duration (24-month follow-up) is justified as it provides sufficient time to observe changes in antibody prevalence over the course of the COVID-19 pandemic as well as sufficient time to determine long term clinical outcomes for pwCF who are SARS-CoV-2 seropositive. Furthermore, we anticipate the 2-year study follow-up period will provide sufficient time to observe the impact of vaccination on antibody levels given that a number of vaccines are now commercially available.

The investigators will compare the level of antibody responses between natural COVID-19 infection and vaccination in pwCF and how this varies over time. This will be achieved by analyzing seroprevalence and antibody levels according to natural infection and vaccination status and according to time of sample post infection or post vaccination, if known.

Optional Study sample collection:

For participants who consent, a second blood sample will also be drawn into EDTA tubes (plasma). Consent to this optional study sample would allow this sample and any remaining serum (following antibody testing) to be stored for future analysis and allow further research to be carried out on related studies to COVID-19 and CF.

ELIGIBILITY:
Inclusion Criteria:

* Consenting people with cystic fibrosis of any age, genotype, transplant status and disease severity.

Exclusion Criteria:

* Refusal to give informed consent
* Contraindication to venepuncture.

Participants already enrolled in a clinical trial are eligible for enrollment in this study. Inclusion in CAR-CF should not preclude enrollment in other observational clinical trial studies or clinical trials of an investigational medicinal product (CTIMP).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consenting people with cystic fibrosis of any age, genotype, transplant status and disease severity will be eligible to participate in the study. The study population is expected to be representative of the general CF population.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
To evaluate SARS-CoV-2 seroprevalence | 3-year period (comprising a 1-year enrollment period and a 2-year follow-up)
  proportion of pwCF with at least 1 seropositive result over the study period and the difference in this proportion by age, geographical area and over time.
To examine the associations | 3-year period (comprising a 1-year enrollment period and a 2-year follow-up)
  Association of SARS-CoV-2 seropositivity, clinical symptoms and clinical outcomes in pwCF: incidence of symptomatic COVID-19 over the study period and severity; proportion of seropositive pwCF with subsequent CF exacerbation compared to pwCF who are seronegative; death rate in pwCF with at least one seropositive result compared to pwCF who are seronegative.
To perform a longitudinal comparison | 3-year period (comprising a 1-year enrollment period and a 2-year follow-up)
  Longitudinal comparison of the detection including level and duration of anti-SARS-CoV-2 antibodies in pwCF following natural infection and SARS-CoV-2 vaccination.

SECONDARY OUTCOMES:
Storage of samples for future analysis | anticipated 5-10 years
  Serum proteomic and genomic responses of pwCF who are SARS-CoV-2 seropositive an seronegative.

CONTACTS AND LOCATIONS:
Overall Officials: Damian Downey, Dr, Study Director — Queen's University, Belfast
Locations (1):
- Erasmus Medical Center Sophia Children's Hospital, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdollahi E, Champredon D, Langley JM, Galvani AP, Moghadas SM. Temporal estimates of case-fatality rate for COVID-19 outbreaks in Canada and the United States. CMAJ. 2020 Jun 22;192(25):E666-E670. doi: 10.1503/cmaj.200711. Epub 2020 May 22. PMID 32444481
- [Background] Stadlbauer D, Amanat F, Chromikova V, Jiang K, Strohmeier S, Arunkumar GA, Tan J, Bhavsar D, Capuano C, Kirkpatrick E, Meade P, Brito RN, Teo C, McMahon M, Simon V, Krammer F. SARS-CoV-2 Seroconversion in Humans: A Detailed Protocol for a Serological Assay, Antigen Production, and Test Setup. Curr Protoc Microbiol. 2020 Jun;57(1):e100. doi: 10.1002/cpmc.100. PMID 32302069
- [Background] Wolfel R, Corman VM, Guggemos W, Seilmaier M, Zange S, Muller MA, Niemeyer D, Jones TC, Vollmar P, Rothe C, Hoelscher M, Bleicker T, Brunink S, Schneider J, Ehmann R, Zwirglmaier K, Drosten C, Wendtner C. Virological assessment of hospitalized patients with COVID-2019. Nature. 2020 May;581(7809):465-469. doi: 10.1038/s41586-020-2196-x. Epub 2020 Apr 1. PMID 32235945
- [Background] Zhao J, Yuan Q, Wang H, Liu W, Liao X, Su Y, Wang X, Yuan J, Li T, Li J, Qian S, Hong C, Wang F, Liu Y, Wang Z, He Q, Li Z, He B, Zhang T, Fu Y, Ge S, Liu L, Zhang J, Xia N, Zhang Z. Antibody Responses to SARS-CoV-2 in Patients With Novel Coronavirus Disease 2019. Clin Infect Dis. 2020 Nov 19;71(16):2027-2034. doi: 10.1093/cid/ciaa344. PMID 32221519
- [Background] Chandrashekar A, Liu J, Martinot AJ, McMahan K, Mercado NB, Peter L, Tostanoski LH, Yu J, Maliga Z, Nekorchuk M, Busman-Sahay K, Terry M, Wrijil LM, Ducat S, Martinez DR, Atyeo C, Fischinger S, Burke JS, Slein MD, Pessaint L, Van Ry A, Greenhouse J, Taylor T, Blade K, Cook A, Finneyfrock B, Brown R, Teow E, Velasco J, Zahn R, Wegmann F, Abbink P, Bondzie EA, Dagotto G, Gebre MS, He X, Jacob-Dolan C, Kordana N, Li Z, Lifton MA, Mahrokhian SH, Maxfield LF, Nityanandam R, Nkolola JP, Schmidt AG, Miller AD, Baric RS, Alter G, Sorger PK, Estes JD, Andersen H, Lewis MG, Barouch DH. SARS-CoV-2 infection protects against rechallenge in rhesus macaques. Science. 2020 Aug 14;369(6505):812-817. doi: 10.1126/science.abc4776. Epub 2020 May 20. PMID 32434946
- [Background] Petherick A. Developing antibody tests for SARS-CoV-2. Lancet. 2020 Apr 4;395(10230):1101-1102. doi: 10.1016/S0140-6736(20)30788-1. No abstract available. PMID 32247384
- [Background] Wang S, Chou TH, Sakhatskyy PV, Huang S, Lawrence JM, Cao H, Huang X, Lu S. Identification of two neutralizing regions on the severe acute respiratory syndrome coronavirus spike glycoprotein produced from the mammalian expression system. J Virol. 2005 Feb;79(3):1906-10. doi: 10.1128/JVI.79.3.1906-1910.2005. PMID 15650214
- [Background] He Y, Zhou Y, Siddiqui P, Jiang S. Inactivated SARS-CoV vaccine elicits high titers of spike protein-specific antibodies that block receptor binding and virus entry. Biochem Biophys Res Commun. 2004 Dec 10;325(2):445-52. doi: 10.1016/j.bbrc.2004.10.052. PMID 15530413
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Coronaviridae Study Group of the International Committee on Taxonomy of Viruses. The species Severe acute respiratory syndrome-related coronavirus: classifying 2019-nCoV and naming it SARS-CoV-2. Nat Microbiol. 2020 Apr;5(4):536-544. doi: 10.1038/s41564-020-0695-z. Epub 2020 Mar 2. PMID 32123347
- [Background] Colombo C, Burgel PR, Gartner S, van Koningsbruggen-Rietschel S, Naehrlich L, Sermet-Gaudelus I, Southern KW. Impact of COVID-19 on people with cystic fibrosis. Lancet Respir Med. 2020 May;8(5):e35-e36. doi: 10.1016/S2213-2600(20)30177-6. Epub 2020 Apr 15. No abstract available. PMID 32304639
- [Background] Cosgriff R, Ahern S, Bell SC, Brownlee K, Burgel PR, Byrnes C, Corvol H, Cheng SY, Elbert A, Faro A, Goss CH, Gulmans V, Marshall BC, McKone E, Middleton PG, Ruseckaite R, Stephenson AL, Carr SB; Global Registry Harmonization Group. A multinational report to characterise SARS-CoV-2 infection in people with cystic fibrosis. J Cyst Fibros. 2020 May;19(3):355-358. doi: 10.1016/j.jcf.2020.04.012. Epub 2020 Apr 25. PMID 32376098
- [Background] Flight WG, Bright-Thomas RJ, Tilston P, Mutton KJ, Guiver M, Morris J, Webb AK, Jones AM. Incidence and clinical impact of respiratory viruses in adults with cystic fibrosis. Thorax. 2014 Mar;69(3):247-53. doi: 10.1136/thoraxjnl-2013-204000. Epub 2013 Oct 14. PMID 24127019
- [Background] Wang EE, Prober CG, Manson B, Corey M, Levison H. Association of respiratory viral infections with pulmonary deterioration in patients with cystic fibrosis. N Engl J Med. 1984 Dec 27;311(26):1653-8. doi: 10.1056/NEJM198412273112602. PMID 6504106
- [Background] Peckham D, McDermott MF, Savic S, Mehta A. COVID-19 meets Cystic Fibrosis: for better or worse? Genes Immun. 2020 Aug;21(4):260-262. doi: 10.1038/s41435-020-0103-y. Epub 2020 Jul 1. PMID 32606316
- [Background] Wat D. Impact of respiratory viral infections on cystic fibrosis. Postgrad Med J. 2003 Apr;79(930):201-3. doi: 10.1136/pmj.79.930.201. PMID 12743335
- [Background] Bucher J, Boelle PY, Hubert D, Lebourgeois M, Stremler N, Durieu I, Bremont F, Deneuville E, Delaisi B, Corvol H, Bassinet L, Grenet D, Remus N, Vodoff MV, Boussaud V, Troussier F, Leruez-Ville M, Treluyer JM, Launay O, Sermet-Gaudelus I. Lessons from a French collaborative case-control study in cystic fibrosis patients during the 2009 A/H1N1 influenza pandemy. BMC Infect Dis. 2016 Feb 1;16:55. doi: 10.1186/s12879-016-1352-2. PMID 26830335
- [Background] Stanton BA, Hampton TH, Ashare A. SARS-CoV-2 (COVID-19) and cystic fibrosis. Am J Physiol Lung Cell Mol Physiol. 2020 Sep 1;319(3):L408-L415. doi: 10.1152/ajplung.00225.2020. Epub 2020 Jul 15. PMID 32668165
- [Background] Berardis S, Verroken A, Vetillart A, Struyf C, Gilbert M, Gruson D, Gohy S. SARS-CoV-2 seroprevalence in a Belgian cohort of patients with cystic fibrosis. J Cyst Fibros. 2020 Nov;19(6):872-874. doi: 10.1016/j.jcf.2020.08.005. Epub 2020 Aug 11. PMID 32828701
- [Background] Farrell PM, Rosenstein BJ, White TB, Accurso FJ, Castellani C, Cutting GR, Durie PR, Legrys VA, Massie J, Parad RB, Rock MJ, Campbell PW 3rd; Cystic Fibrosis Foundation. Guidelines for diagnosis of cystic fibrosis in newborns through older adults: Cystic Fibrosis Foundation consensus report. J Pediatr. 2008 Aug;153(2):S4-S14. doi: 10.1016/j.jpeds.2008.05.005. PMID 18639722
- [Background] Howie SR. Blood sample volumes in child health research: review of safe limits. Bull World Health Organ. 2011 Jan 1;89(1):46-53. doi: 10.2471/BLT.10.080010. Epub 2010 Sep 10. PMID 21346890
- See also: European Centre for Disease Prevention and Control. Immune responses and immunity to SARS-CoV-2. Published 2020. — https://www.ecdc.europa.eu/en/covid-19/latest-evidence/immune-responses